CLINICAL TRIAL: NCT03966729
Title: Retrospektive Datenanalyse Von Herzinsuffizienzpatienten in Der Kardiologie Des Universitätsklinikums Würzburg
Brief Title: Relationships and Differences Analysis in Heart Failure
Acronym: REDEAL-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, PD Dr. Peter Nordbeck, Head Consultant Cardiology, Wuerzburg University Hospital
Other Study IDs: REDEAL-HF
Record Dates: First submitted 2019-02-04; First posted 2019-05-29 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure; Chronic Heart Failure; Chronic Heart Disease
Keywords: HFmrEF; HFrEF; HFpEF; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFrEF: HFrEF (Heart failure with reduced ejection fraction): ESC Guideline heart failure 2016: patients with LVEF < 40%.
  LVEF = Left ventricular ejection fraction
  Interventions: Other: Time (outcome)
- HFmrEF: HFmrEF (Heart failure with mid-range reduced ejection fraction): ESC Guideline heart failure 2016: patients with LVEF 40-49%.
  LVEF = Left ventricular ejection fraction
  Interventions: Other: Time (outcome)
- HFpEF: HFmrEF (Heart failure with preserved ejection fraction): ESC Guideline heart failure 2016: patients with LVEF > 50%.
  LVEF = Left ventricular ejection fraction
  Interventions: Other: Time (outcome)

INTERVENTIONS:
Other: Time (outcome)

SUMMARY:
This study characterizes heart failure patients who attended the University Hospital Würzburg. The primary aim is a better understanding of the relationships and differences between the subgroups HFrEF (EF < 40%), HFmrEF (EF 40-49%), and HFpEF (EF>50%), contributing to an improved diagnosis, prognosis and therapy of patients with heart failure.

DETAILED DESCRIPTION:
The varying clinical picture of heart failure (HF) represents a major challenge for patient care in Germany. HF is one of the most common reasons for hospitalization in the Western world. In the chronic course of heart failure, affected patients are committed to morbidity, lifelong therapy and high risk of cardiac decompensation, also associated with high mortality.

Heart failure patients, who visited the Cardiology Department of the University Hospital Wuerzburg, shall be analyzed with regard to all clinical data and outcome. This retrospective work should help to better understand the three groups HFrEF (EF < 40%), HFmrEF (EF 40-49%) and HFpEF (EF>50%) and help identifying similarities and differences between the groups.

Hereby we hope for progress in diagnostic, prognostic and therapeutic aspects of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Heart failure
* Minimum of two echocardiographic examinations in a minimum time frame of six months
* Patients must have reached the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our cohort consists of patients who attended the Cardiology Department of University Hospital Wuerzburg in the time period between 2009 and 2019.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term survival in heart failure patients with preserved, mid-range or reduced left ventricular ejection fraction | 1 year follow up after last examination
  Survival of patients with heart failure extracted from medical record or by telephone interview

SECONDARY OUTCOMES:
Impact of clinical imaging and laboratory parameters on long-term survival in heart failure patients with precerved, mid-range or reduced left ventricular ejection fraction | 6 months
  Parameters are derived from standard echocardiography, cardiac magnetic resonance imaging and blood testing.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nordbeck, MD, PhD, Study Chair — Wuerzburg University Hospital
Locations (1):
- University Hospital Würzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No